CLINICAL TRIAL: NCT01847443
Title: A Pharmacokinetic Study Comparing Two Nicotine Gum Formulations in a Single Dose Design
Brief Title: Comparison of Pharmacokinetic Profiles of Two Nicotine Gum Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RH01705
Record Dates: First submitted 2013-05-02; First posted 2013-05-06 (Estimated); Results first posted 2014-04-11 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-01

CONDITIONS: Smoking Cessation
Keywords: nicotine; nicotine replacement therapy; nicotine gum
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test nicotine gum (2 mg) (Experimental): A single dose of Nicotine Mint Gum (2 mg) to be chewed.
  Interventions: Drug: Nicotine (2 mg)
- Test nicotine gum (4 mg) (Experimental): A single dose of Nicotine Mint Gum (4 mg) to be chewed.
  Interventions: Drug: Nicotine (4 mg)
- Reference nicotine gum (2 mg) (Active Comparator): A single dose of reference nicotine gum (2 mg) to be chewed.
  Interventions: Drug: Nicotine (2 mg)
- Reference nicotine gum (4 mg) (Active Comparator): A single dose of reference nicotine gum (4 mg) to be chewed.
  Interventions: Drug: Nicotine (4 mg)

INTERVENTIONS:
Drug: Nicotine (2 mg) — 2 mg nicotine gum in two formulations
  Arms: Reference nicotine gum (2 mg); Test nicotine gum (2 mg)
Drug: Nicotine (4 mg) — 4 mg nicotine gum in two formulations
  Arms: Reference nicotine gum (4 mg); Test nicotine gum (4 mg)

SUMMARY:
The primary objective of this study is to compare pharmacokinetic (PK) profiles and assess the bioequivalence between the newly developed nicotine gums (2 mg and 4 mg) and the reference nicotine gums (2 mg and 4 mg) in healthy smokers.

ELIGIBILITY:
Inclusion Criteria:

* BMI within the range of 19 to 30 kilograms/meters^2
* Current cigarette smokers who have smoked daily for at least a year, and smoke their first cigarette within 30 minutes of waking up

Exclusion Criteria:

* Participants who have attempted to quit smoking in the last 12 months, are currently attempting to quit smoking or reduce the number of cigarettes they smoke, or are intending to quit smoking in the next 3 months, with or without use of smoking cessation aids
* Treatment with known hepatic enzyme altering agents

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Celerion - BELFAST, Belfast, Northern Ireland, United Kingdom

REFERENCES:
- [Derived] Du D. A Single-Dose, Crossover-Design Bioequivalence Study Comparing Two Nicotine Gum Formulations in Healthy Subjects. Adv Ther. 2018 Aug;35(8):1169-1180. doi: 10.1007/s12325-018-0752-7. Epub 2018 Jul 19. PMID 30027479

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were recruited at a single site in the UK.
Pre-assignment Details: A total of 160 participants were screened for this study, of which 84 participants were randomized. Seventy seven participants completed the study.
Groups:
- 2mg Mint Gum/4mg Ref Gum/4mg Mint Gum/2mg Ref Gum: Participants randomly received 2mg nicotine mint gum or 4mg reference (ref) nicotine gum or 4mg nicotine mint gum or 2mg ref nicotine gum once daily on Day 1 of treatment period 1. After a 2-7 day washout period, participants were returned to the next treatment period until all four treatment periods were completed.
- 4mg Ref Gum/2mg Ref Gum/2mg Mint Gum/4mg Mint Gum: Participants randomly received 4mg ref nicotine gum or 2mg ref nicotine gum or 2mg nicotine mint gum or 4mg nicotine mint gum once daily on Day 1 of treatment period 1. After a 2-7 day washout period, participants were returned to the next treatment period until all four treatment periods were completed.
- 2mg Ref Gum/4mg Mint Gum/4mg Ref Gum/2mg Mint Gum: Participants randomly received 2mg ref nicotine gum or 4mg nicotine mint gum or 4mg ref nicotine gum or 2mg nicotine mint gum once daily on Day 1 of treatment period 1. After a 2-7 day washout period, participants were returned to the next treatment period until all four treatment periods were completed.
- 4mg Mint Gum/2mg Mint Gum/2mg Ref Gum/4mg Ref Gum: Participants randomly received 4mg nicotine mint gum or 2mg nicotine mint gum or 2mg ref nicotine gum or 4mg ref nicotine gum once daily on Day 1 of treatment period 1. After a 2-7 day washout period, participants were returned to the next treatment period until all four treatment periods were completed.
Period: Study Period 1
Arm/Group | 2mg Mint Gum/4mg Ref Gum/4mg Mint Gum/2mg Ref Gum | 4mg Ref Gum/2mg Ref Gum/2mg Mint Gum/4mg Mint Gum | 2mg Ref Gum/4mg Mint Gum/4mg Ref Gum/2mg Mint Gum | 4mg Mint Gum/2mg Mint Gum/2mg Ref Gum/4mg Ref Gum
Started | 21 | 21 | 21 | 21
Completed | 21 | 20 | 21 | 21
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Washout Period Before Study Period 2
Arm/Group | 2mg Mint Gum/4mg Ref Gum/4mg Mint Gum/2mg Ref Gum | 4mg Ref Gum/2mg Ref Gum/2mg Mint Gum/4mg Mint Gum | 2mg Ref Gum/4mg Mint Gum/4mg Ref Gum/2mg Mint Gum | 4mg Mint Gum/2mg Mint Gum/2mg Ref Gum/4mg Ref Gum
Started | 21 | 20 | 21 | 21
Completed | 19 | 19 | 21 | 21
Not Completed | 2 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Other reason | 1 | 0 | 0 | 0
Period: Study Period 2
Arm/Group | 2mg Mint Gum/4mg Ref Gum/4mg Mint Gum/2mg Ref Gum | 4mg Ref Gum/2mg Ref Gum/2mg Mint Gum/4mg Mint Gum | 2mg Ref Gum/4mg Mint Gum/4mg Ref Gum/2mg Mint Gum | 4mg Mint Gum/2mg Mint Gum/2mg Ref Gum/4mg Ref Gum
Started | 19 | 19 | 21 | 21
Completed | 19 | 19 | 21 | 21
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period Before Study Period 3
Arm/Group | 2mg Mint Gum/4mg Ref Gum/4mg Mint Gum/2mg Ref Gum | 4mg Ref Gum/2mg Ref Gum/2mg Mint Gum/4mg Mint Gum | 2mg Ref Gum/4mg Mint Gum/4mg Ref Gum/2mg Mint Gum | 4mg Mint Gum/2mg Mint Gum/2mg Ref Gum/4mg Ref Gum
Started | 19 | 19 | 21 | 21
Completed | 18 | 19 | 21 | 21
Not Completed | 1 | 0 | 0 | 0
Not completed — Other reason | 1 | 0 | 0 | 0
Period: Study Period 3
Arm/Group | 2mg Mint Gum/4mg Ref Gum/4mg Mint Gum/2mg Ref Gum | 4mg Ref Gum/2mg Ref Gum/2mg Mint Gum/4mg Mint Gum | 2mg Ref Gum/4mg Mint Gum/4mg Ref Gum/2mg Mint Gum | 4mg Mint Gum/2mg Mint Gum/2mg Ref Gum/4mg Ref Gum
Started | 18 | 19 | 21 | 21
Completed | 18 | 19 | 21 | 21
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period Before Study Period 4
Arm/Group | 2mg Mint Gum/4mg Ref Gum/4mg Mint Gum/2mg Ref Gum | 4mg Ref Gum/2mg Ref Gum/2mg Mint Gum/4mg Mint Gum | 2mg Ref Gum/4mg Mint Gum/4mg Ref Gum/2mg Mint Gum | 4mg Mint Gum/2mg Mint Gum/2mg Ref Gum/4mg Ref Gum
Started | 18 | 19 | 21 | 21
Completed | 16 | 19 | 21 | 21
Not Completed | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Positive alcohol test | 1 | 0 | 0 | 0
Period: Study Period 4
Arm/Group | 2mg Mint Gum/4mg Ref Gum/4mg Mint Gum/2mg Ref Gum | 4mg Ref Gum/2mg Ref Gum/2mg Mint Gum/4mg Mint Gum | 2mg Ref Gum/4mg Mint Gum/4mg Ref Gum/2mg Mint Gum | 4mg Mint Gum/2mg Mint Gum/2mg Ref Gum/4mg Ref Gum
Started | 16 | 19 | 21 | 21
Completed | 16 | 19 | 21 | 21
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Participants
Number analyzed (Participants) | 84
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.8 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 44

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time 0 to Time 't' [AUC(0-t)] of Nicotine 2 mg Test and Reference Product
Description: AUC(0-t) for 2 mg test was compared with 2 mg reference gum
Time Frame: Blood samples to be collected from baseline to 12 hours post dose
Population: Bioequivalence evaluable subjects' population: participants randomized to 1 of 4 treatment sequences; took atleast one dose of study medication (both test and reference) in 2 mg dose and/or in 4 mg doses; did not have any adverse event assimilated to vomiting in first 4 h post-treatment; and did not have baseline nicotine concentration >5% of Cmax.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Test Nicotine Gum (2 mg) | Reference Nicotine Gum (2 mg)
Number analyzed (Participants) | 62 | 62
hr*ng/mL | 11.49 (4.224) | 10.24 (3.768)
Statistical Analysis 1: Comparison: Test Nicotine Gum (2 mg) vs Reference Nicotine Gum (2 mg); Null hypothesis stated that there was no difference between the test and reference gums in AUC(0-t); Test type: Non-Inferiority or Equivalence — Bioequivalence was to be established between the test and reference treatment if the 90% CI of ratio of geometric means (Test/Reference) was included within the bioequivalence limits of (0.80, 1.25); ANOVA; Ratio of Geometric means = 1.107, 90% CI 2-sided [1.070 to 1.147]

2. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Nicotine 2 mg Test and Reference Products, and Nicotine 4 mg Test and Reference Products
Description: Tmax for 2 mg test was compared with 2 mg reference gum, and 4 mg test was compared with 4 mg reference gum
Time Frame: Blood samples to be collected from baseline to 12 hours post dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Test Nicotine Gum (2 mg) | Reference Nicotine Gum (2 mg) | Test Nicotine Gum (4 mg) | Reference Nicotine Gum (4 mg)
Number analyzed (Participants) | 62 | 62 | 73 | 73
hr | 0.75 [0.5 to 1.0] | 0.75 [0.5 to 1.5] | 0.75 [0.5 to 1.5] | 0.75 [0.2 to 2.0]

3. Secondary Outcome: Apparent Terminal Elimination Half-life (T1/2) of Nicotine 2 mg Test and Reference Products, and Nicotine 4 mg Test and Reference Products
Description: T1/2 of 2 mg test was compared with 2 mg reference gum, and 4 mg test was compared with 4 mg reference gum
Time Frame: Blood samples to be collected from baseline to 12 hours post dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Test Nicotine Gum (2 mg) | Reference Nicotine Gum (2 mg) | Test Nicotine Gum (4 mg) | Reference Nicotine Gum (4 mg)
Number analyzed (Participants) | 62 | 62 | 73 | 73
hr | 2.12 [1.4 to 3.4] | 2.03 [1.2 to 4.2] | 2.01 [1.3 to 4.1] | 2.02 [1.3 to 3.4]

4. Secondary Outcome: Apparent Terminal Elimination Rate Constant (Kel) of Nicotine 2 mg Test and Reference Products, and Nicotine 4 mg Test and Reference Products
Description: Kel for 2 mg test was compared with 2 mg reference gum, and 4 mg test was compared with 4 mg reference gum
Time Frame: Blood samples to be collected from baseline to 12 hours post dose
Population: as for outcome 1
Measure: Median (Full Range); unit: 1/hr
Arm/Group | Test Nicotine Gum (2 mg) | Reference Nicotine Gum (2 mg) | Test Nicotine Gum (4 mg) | Reference Nicotine Gum (4 mg)
Number analyzed (Participants) | 62 | 62 | 73 | 73
1/hr | 0.33 [0.2 to 0.5] | 0.34 [0.2 to 0.6] | 0.34 [0.2 to 0.5] | 0.34 [0.2 to 0.5]

5. Secondary Outcome: Area Under Concentration-time Curve From Time 0 Extrapolated to ∞ [AUC(0-∞)] of Nicotine 2 mg Test and Reference Products, and Nicotine 4 mg Test and Reference Products
Description: AUC(0-∞) for 2mg test was compared with 2 mg reference gum, and 4 mg test was compared with 4 mg reference gum
Time Frame: Blood samples to be collected from baseline to 12 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Test Nicotine Gum (2 mg) | Reference Nicotine Gum (2 mg) | Test Nicotine Gum (4 mg) | Reference Nicotine Gum (4 mg)
Number analyzed (Participants) | 62 | 62 | 73 | 73
hr*ng/mL | 12.56 (4.409) | 11.20 (3.955) | 24.60 (7.845) | 22.64 (7.136)

6. Primary Outcome: AUC(0-t) of Nicotine 4 mg Test and Reference Product
Description: AUC(0-t) of Nicotine 4 mg test was compared with 4 mg reference gum
Time Frame: Blood samples to be collected from baseline to 12 hours post dose
Population: Bioequivalence evaluable subjects' population: participants randomized to 1of 4 treatment sequences; took atleast one dose of study medication (both test and ref) in 2 mg dose and/or in 4 mg doses; did not have any AE assimilated to vomiting in first 4h post-treatment; and did not have baseline nicotine concentration >5% of Cmax.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Test Nicotine Gum (4 mg) | Reference Nicotine Gum (4 mg)
Number analyzed (Participants) | 73 | 73
hr*ng/mL | 23.44 (7.593) | 21.50 (6.874)
Statistical Analysis 1: Comparison: Test Nicotine Gum (4 mg) vs Reference Nicotine Gum (4 mg); Null hypothesis stated that there was no difference between the test and reference gums in AUC(0-t); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of Geometric means = 1.098, 90% CI 2-sided [1.061 to 1.137]

7. Primary Outcome: Maximum Observed Concentration (Cmax) of Nicotine 2 mg Test and Reference Product
Description: Cmax for 2 mg test was compared with 2 mg reference gum
Time Frame: Blood samples to be collected from baseline to 12 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Test Nicotine Gum (2 mg) | Reference Nicotine Gum (2 mg)
Number analyzed (Participants) | 62 | 62
ng/mL | 3.93 (1.232) | 3.72 (1.289)
Statistical Analysis 1: Comparison: Test Nicotine Gum (2 mg) vs Reference Nicotine Gum (2 mg); Null hypothesis stated that there was no difference between the test and reference gums in Cmax; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of Geometric means = 1.044, 90% CI 2-sided [1.002 to 1.089]

8. Primary Outcome: Cmax of Nicotine 4 mg Test and Reference Product
Description: Cmax for 4 mg test was compared with 4 mg reference gum
Time Frame: Blood samples to be collected from baseline to 12 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Test Nicotine Gum (4 mg) | Reference Nicotine Gum (4 mg)
Number analyzed (Participants) | 73 | 73
ng/mL | 7.49 (1.720) | 6.98 (1.777)
Statistical Analysis 1: Comparison: Test Nicotine Gum (4 mg) vs Reference Nicotine Gum (4 mg); Null hypothesis stated that there was no difference between the test and reference gums in Cmax; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of Geometric means = 1.071, 90% CI 2-sided [1.028 to 1.116]

ADVERSE EVENTS:
Arm/Group | Test Nicotine Gum (2 mg) | Reference Nicotine Gum (2 mg) | Test Nicotine Gum (4 mg) | Reference Nicotine Gum (4 mg)
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/77 | 0/79 | 0/81
Other Adverse Events (participants affected / at risk) | 11/82 | 12/77 | 12/79 | 11/81
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Nicotine Gum (2 mg) (N=82) | Reference Nicotine Gum (2 mg) (N=77) | Test Nicotine Gum (4 mg) (N=79) | Reference Nicotine Gum (4 mg) (N=81)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Catheter site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site anaesthesia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vessel puncture site pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 4 (4) | 5 (5) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.